CLINICAL TRIAL: NCT02104089
Title: Post-market Observational Study Zenith® t-Branch™ Thoracoabdominal Endovascular Graft
Brief Title: Post-market Observational Study Zenith® t-Branch™
Status: Completed | Type: Observational
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-017
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Aortic Aneurysm; Thoracoabdominal
Keywords: Thoracoabdominal aortic aneurysm; Endovascular; Fenestration; Branch; Off-the-shelf
MeSH Terms: conditions — Aortic Aneurysm; Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other

GROUPS / COHORTS (1):
- Endovascular treatment: Zenith® t-Branch™ Thoracoabdominal Endovascular Graft
  Interventions: Device: Zenith® t-Branch™ Thoracoabdominal Endovascular Graft

INTERVENTIONS:
Device: Zenith® t-Branch™ Thoracoabdominal Endovascular Graft — Instead of making a large incision in the chest, the physician makes a small incision near each hip to insert, and guide the study device(s) into place in the aorta.

SUMMARY:
The Zenith® t-Branch™ Thoracoabdominal Endovascular Graft Study is a post-market observational study to evaluate the performance of the Zenith® t-Branch™ in the treatment of thoracoabdominal aortic aneurysms in routine care.

DETAILED DESCRIPTION:
Both retrospective and prospective patients will be enrolled

ELIGIBILITY:
Inclusion Criteria:

* Treated with the off-the-shelf Zenith® t-Branch™ Thoracoabdominal Endovascular Graft
* Signed informed consent

Exclusion Criteria:

* Inability or refusal to give informed consent by the patient or a legally authorized representative

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
Rate of mortality and morbidity | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni B Torsello, M.D., Principal Investigator — St. Franziscus Hospital-GmbH
Locations (3):
- Germany (2):
  - Universitäts Krankenhaus Eppendorf, Hamburg
  - St. Franziscus Hospital-GmbH, Münster
- Skaane University Hospital, Malmo, Sweden

REFERENCES:
- [Derived] Tsilimparis N, Bosiers M, Resch T, Torsello G, Austermann M, Rohlffs F, Coates B, Yeh C, Kolbel T. Two-year target vessel-related outcomes following use of off-the-shelf branched endografts for the treatment of thoracoabdominal aortic aneurysms. J Vasc Surg. 2023 Aug;78(2):289-298. doi: 10.1016/j.jvs.2023.03.498. Epub 2023 Apr 11. PMID 37044318
- [Derived] Bosiers M, Kolbel T, Resch T, Tsilimparis N, Torsello G, Austermann M. Early and midterm results from a postmarket observational study of Zenith t-Branch thoracoabdominal endovascular graft. J Vasc Surg. 2021 Oct;74(4):1081-1089.e3. doi: 10.1016/j.jvs.2021.01.070. Epub 2021 Mar 5. PMID 33684474